CLINICAL TRIAL: NCT06435858
Title: Short-term Effects of an SGLT2 Inhibitor on Divalent Ions in Autosomal Dominant Polycystic Kidney Disease
Acronym: SIDIA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cantonal Hospital Graubuenden (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, Patrick Hofmann, Principal Investigator, Cantonal Hospital Graubuenden
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-00070
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-03

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: phosphate; calcium; magnesium; Empagliflozin; ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Investigator-initiated randomised, single-blind, placebo-controlled, cross-over study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Empagliflozin 10mg
  Interventions: Drug: Empagliflozin
- Control (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin 10mg
  Arms: Intervention
Drug: Placebo — Placebo capsule
  Arms: Control

SUMMARY:
This study aims to better understand electrolyte handling in patients with autosomal dominant polycystic kidney disease treated with the SGLT2 inhibitor Empagliflozin.

Patients will be randomized into two groups and take Empagliflozin or a Placebo for 2 weeks with a wash-out period of 2 weeks. The primary outcome is tubular handling of the divalent ions calcium, phosphate and magnesium. Secondary outcomes include diuresis, safety and tolerability.

DETAILED DESCRIPTION:
This investigator-initiated randomised, single-blind, placebo-controlled cross-over study aims to better understand tubular electrolyte handling of divalent ions in patients with autosomal dominant polycystic kidney disease treated with the SGLT2 inhibitor Empagliflozin.

After randomization, at week 0, participants collect 24-hour urine sample and a patient visit to assess vitals and blood tests takes place. After this visit, period 1 starts with a 2-week treatment of either Empagliflozin 10mg or Placebo.

At week 2, the second 24-hour-urine sample and 2. patient visit and blood test take place. After this visit, wash-out period for 2 weeks starts where no study drug will be administered At week 4, the period 2, the crossover-period starts for an additional 2 weeks. At week 6; a final and third 24-hour urine sample, clinical visit and blood test takes place.

At week 3 & 7, a phone consultation will assess safety.

ELIGIBILITY:
Inclusion Criteria:

* - Patients 18-75 years old with ADPKD, defined according to international diagnostic and classification criteria14, treated at Cantonal Hospital Graubünden (KSGR) and the University Hospital Zürich (USZ) independent of baseline treatment with the vasopressin receptor antagonist Tolvaptan
* Informed consent as documented by signature

Exclusion Criteria:

* - renal replacement therapy or kidney allograft recipient
* chronic kidney disease CKD KDIGO Stage G4 (eGFR under 30ml/min/1.73m2)
* patients younger 18 years of age
* Diabetes mellitus type 1
* recurrent urinary tract infections (UTI) defined as more than 3 infections requiring antibiotic treatment or over 1 requiring hospitalization/year.
* Patients with uncontrolled hypertension (defined as ambulatory systolic BP over 180mmHg), liver cirrhosis (Child Pugh B and C)
* Patients not able or not willing to stop the following medications during the study period of participation in the trial:
* Thiazide diuretics
* Carbonic anhydrase inhibitors
* Sodium bicarbonate
* 1, 25 (OH) vitamin D (calcitriol)
* Bisphosphonate, denosumab, teriparatide
* Pregnant or lactating women
* Known allergy to study drug
* Inability to understand and follow the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | After a two week intervention
  - Calcium, phosphate, magnesium excretion

SECONDARY OUTCOMES:
Secondary Outcome | After a two week intervention
  - diuresis (24-hour urine volume, 24-hour creatinine, ketonuria, osmolarity, urinary pH) - tubular handling of other electrolytes (Na, K, Cl) - inflammation metabolism (CRP, hemoglobin?) - kidney function (creatinine, uric acid, urea, hemoglobin?) - effect on standardized blood pressure (assessed every two weeks) - bone metabolism (FGF23, PTH, 25-(OH)-D3) - tolerability (patient-reported side effects (nycturia, urinary urgency, lightheadedness, syncope) - safety (bacteriuria, urinary tract infection requiring antibiotic treatment, genital mycosis)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Fehr, MD, Principal Investigator — Cantonal Hospital Graubuenden; Patrick Hofmann, MD, Principal Investigator — Cantonal Hospital Graubuenden
Locations (2):
- Switzerland (2):
  - University Hospital Zurich, Division of Nephrology, Zurich, Canton of Zurich
  - Cantonal Hospital Graubuenden, Chur, Kanton Graubünden

IPD SHARING:
Plan to Share IPD: No
The local ethics committee approval does not include individual participant data sharing.

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039